CLINICAL TRIAL: NCT02431442
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RM 493 Administered to Healthy Obese Non-diabetic Volunteers
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RM-493 Administered to Healthy, Obese, Non-diabetic Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RM-493-002
Record Dates: First submitted 2015-04-22; First posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Overweight; Obese
Keywords: Heterozygous; MC4R deficiency; associated
MeSH Terms: conditions — Overweight; Obesity | interventions — setmelanotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (12):
- Cohort 1: RM-493 SC Infusion 14 Days (Active Comparator): Double-blind RM-493 will be administered at a dose of 0.01 mg/kg/24 hours via subcutaneous continuous infusion for 14 days (1 panel, all male subjects)
  Interventions: Drug: RM-493
- Cohort 2: RM-493 SC Infusion 28 Days (Active Comparator): Double-blind RM-493 will be administered at a dose of 0.01 mg/kg/24 hours via subcutaneous continuous infusion for 28 days (1 panel)
  Interventions: Drug: RM-493
- Cohort 3: RM-493 SC Infusion 28 Days (Active Comparator): Double-blind RM-493 will be administered at a dose of 0.01 mg/kg/24 hours via subcutaneous continuous infusion for 28 days (1 panel)
  Interventions: Drug: RM-493
- Cohort 4: RM-493 SC Infusion 28 Days (Active Comparator): Double-blind RM-493 will be administered at a dose of 0.015 mg/kg/24 hours via subcutaneous continuous infusion for 28 days (1 panel)
  Interventions: Drug: RM-493
- Cohort 5: RM-493 SC Injection 14 days (Active Comparator): Double-blind RM-493 will be administered at a dose of 0.0075 mg/kg every 12 hours via a subcutaneous injection for 14 days (1 panel)
  Interventions: Drug: RM-493
- Cohort 6: RM-493 SC Infusion 28 Days (Active Comparator): Double-blind RM-493 will be administered at a dose of 0.01 mg/kg/24 hours via subcutaneous continuous infusion for 28 days (1 panel, heterozygous MC4R subjects)
  Interventions: Drug: RM-493
- Cohort 1: Placebo SC Infusion 14 Days (Placebo Comparator): Double-blind Placebo will be administered via subcutaneous continuous infusion for 14 days (1 panel, all male subject)
  Interventions: Drug: Placebo
- Cohort 2: Placebo SC Infusion 28 Days (Placebo Comparator): Double-blind Placebo will be via subcutaneous continuous infusion for 14 days (1 panel)
  Interventions: Drug: Placebo
- Cohort 3: Placebo SC Infusion 28 Days (Placebo Comparator): Double-blind Placebo will be administered via subcutaneous continuous infusion for 28 days (1 panel)
  Interventions: Drug: Placebo
- Cohort 4: Placebo SC Infusion 28 Days (Placebo Comparator): Double-blind Placebo will be administered via subcutaneous continuous infusion for 28 days (1 panel)
  Interventions: Drug: Placebo
- Cohort 5: Placebo SC Injection 14 days (Placebo Comparator): Double-blind Placebo will be administered via a subcutaneous injection every 12 hours for 14 days (1 panel)
  Interventions: Drug: Placebo
- Cohort 6: Placebo SC Infusion 28 Days (Placebo Comparator): Double-blind Placebo will be administered via subcutaneous continuous infusion for 28 days (1 panel, heterozygous MC4R subjects)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RM-493
  Other Names: setmelanotide
  Arms: Cohort 1: RM-493 SC Infusion 14 Days; Cohort 2: RM-493 SC Infusion 28 Days; Cohort 3: RM-493 SC Infusion 28 Days; Cohort 4: RM-493 SC Infusion 28 Days; Cohort 5: RM-493 SC Injection 14 days; Cohort 6: RM-493 SC Infusion 28 Days
Drug: Placebo
  Arms: Cohort 1: Placebo SC Infusion 14 Days; Cohort 2: Placebo SC Infusion 28 Days; Cohort 3: Placebo SC Infusion 28 Days; Cohort 4: Placebo SC Infusion 28 Days; Cohort 5: Placebo SC Injection 14 days; Cohort 6: Placebo SC Infusion 28 Days

SUMMARY:
The purpose of this study is to evaluate the multiple dose safety and tolerability of RM-493 (setmelanotide) as well as pharmacokinetic (PK) and pharmacodynamic (PD; weight loss) profile, in healthy obese patients for 2 to 4 weeks. In addition, one panel of patients with a specific genetic deficiency in the hypothalamic leptin- proopiomelanocortin (POMC) - melanocortin-4 receptor (MC4R) pathway, those with heterozygous partial or full loss of function (LOF) of the MC4R gene, will also be studied. The study drug (RM-493 and placebo) will be administered subcutaneously in a blinded fashion by subcutaneous (SC) infusion or injection.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide voluntary, written informed consent with comprehension of all aspects of the protocol, prior to any study procedures.
* Healthy obese male and female volunteers aged 18 to 55 years, inclusive. Heterozygous subjects may be 18 to 65 years inclusive.
* In good general health, without significant medical history, physical examination findings, or clinical laboratory abnormalities.
* Body Mass Index of 30-40 kg/m2, inclusive. Heterozygous subjects may have a broader BMI range; to be eligible heterozygous subjects may have a BMI 27 -55 kg/ m2, inclusive.
* Stable body weight during the previous 6 months, based on Investigator judgment.
* Blood pressure <140/90 mmHg at Screening and D-1. Measurement may be repeated within 24 hours, based on Investigator judgment.
* Females must not be pregnant and must have a negative serum pregnancy test result at the Screening Visit and Day -1.
* Females of childbearing potential must agree to be abstinent or else use any two of the following medically acceptable forms of contraception from the Screening Period through the Final Study Visit: hormonal, condom with spermicidal jelly, diaphragm or cervical cap with spermicidal jelly, or IUD. Hormonal contraception must have started at least 3 months prior to screening. A female whose male partner has had a vasectomy must agree to use one additional form of medically acceptable contraception. Subjects must agree to practice the above birth control methods for 30 days from the final visit as a safety precaution.
* Females of non-childbearing potential, defined as surgically sterile (status post hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or post-menopausal for at least 12 months (and confirmed with a screening FSH level in the post-menopausal range), do not require contraception during the study.
* Males with female partners of childbearing potential must agree to use two medically acceptable forms of contraception as described above, with one of the two forms being condom with spermicide, from the Screening Period through the Final Study Visit. Males with female partners of childbearing potential who themselves are surgically sterile (status post vasectomy) must agree to use condoms with spermicide over the same period of time. Male subjects must agree to practice the above birth control methods for 30 days from the final visit as a safety precaution.

Exclusion Criteria:

* Fasting blood glucose >126 mg/dL at screening. Heterozygous subjects will be excluded for a fasting blood glucose >140 mg/dL.
* Resting heart rate <45 bpm or >90 bpm at screening.
* Abnormal thyroid stimulating hormone (TSH) or thyroxine (T4) levels on screening.
* Elevated ALT or serum creatinine on screening or any clinically significant abnormalities on screening laboratory tests as determined by the Investigator.
* History of medically treated diabetes or of treated or medically diagnosed hypertension. Heterozygous subjects who have diagnosed hypertension and are well controlled on treatment (Refer to Exclusion Criteria 20 below), are eligible. .
* Presence of a skin lesion suspicious for malignancy, unless excised prior to Day 1.
* History of malignancy except for treated cervical carcinoma in situ in the past 5 years.
* Active or history of any clinically significant medical condition including renal, hepatic, pulmonary, gastrointestinal, cardiovascular, genitourinary, endocrine, immunologic, metabolic, neurologic, psychiatric or hematological disease, based on Investigator judgment.
* Acute illness or history of illness, which in the opinion of the Investigator, could pose a threat or harm to the subject or obscure interpretation of laboratory test results or interpretation of study data.
* Positive hepatitis B surface antigen, positive hepatitis C antibody or positive HIV test at screening or a history of positive testing (e.g. liver biopsy, serology) suggesting acute or chronic hepatitis.
* Abnormal 12-lead electrocardiogram (ECG) at screening or pre-dose (Day -1 or Day 1), except minor deviations deemed to be of no clinical significance by the Investigator.
* Received any experimental drugs or devices within 30 days or 5 half lives, whichever is longer, prior to dosing.
* Ongoing participation in a prior clinical study at the time of screening.
* Blood donation within 60 days prior to screening or intent to donate within 60 days after Final Study Visit.
* Hospitalization for major surgery including but not limited to abdominal, thoracic, or cardiovascular surgery within the past 3 months prior to screening, or for a clinically significant non-surgical illness, based on Investigator judgment, within the past 3 months.
* Planned elective surgery within 30 days of the Final Study Visit.
* Poor venous access or inability to tolerate venipuncture.
* History of significant drug hypersensitivity or anaphylaxis.
* History of hypersensitivity to proteins (e.g., allergy shots).
* Use of prescription medications on a regular basis. The last use of any prescription medication must have been greater than 5 half-lives for the specific medication or at least 14 days prior to admission (Day -1), whichever is longer. Hormonal contraception is allowed for female subjects.

Heterozygous cohorts: Use of prescription medications on a regular basis is not allowed with the following exceptions:

* Antihypertensives (<3 medications on a stable dose for ≥ 30 days);
* Statins (dose must be ≤ half the maximum dose; must be on a stable dose ≥3 months);
* Fibrates (must be on stable dose for ≥3 months);
* Niacin (must be on stable dose for ≥3 months);
* Thyroxin (stable dose for ≥ 30 days); The last use of any other prescription medication will need follow the criteria for all other cohorts, as outlined above.

Use of prescription medications not listed above may be allowed at the discretion of the Investigator upon consultation with Rhythm.

* Use of a non-prescription drug and herbal substances during the study (through the Final Study Visit). The last dose of any non-prescription drug must have been taken greater than 5 half-lives for that drug before receiving study drug.
* Inability to attend all study visits or to comply with protocol requirements including fasting and restrictions on alcohol, caffeine, nicotine and concomitant medication intake.
* A significant history of drug/solvent abuse within 5 years of screening or a positive test for drugs of abuse test at screening or on Day -1.
* Positive alcohol (breath test) or nicotine screen at Screening Visit or Day 1 (positive nicotine screen does not apply to heterozygous cohort).
* History of alcohol abuse (defined as average intake of three or more units of alcohol per day) within 5 years of the Screening Visit.
* History of tobacco or tobacco product use unless abstinent for at least one year prior to the Screening Visit. This criterion does not apply to heterozygous subjects.
* Previously randomized and dosed in this study. This criterion does not apply to heterozygous subjects.
* Any other reason, which in the opinion of the Investigator would confound proper evaluation of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of adverse events. | Day 1 through Day 14 or Day 28 (depending on Cohort)

SECONDARY OUTCOMES:
Pharmacokinetics (PK) Profile | Day 1 through Day 14 or Day 28 (depending on Cohort)
  Frequent PK (trough) sampling throughout the study, including 24-hour inpatient PK profiles at the beginning and end of the study.
Assessment of weight loss based on weight measurements | Day 1 through Day 14 or Day 28 (depending on Cohort)
Assessment of blood pressure using Ambulatory blood pressure monitors. | Day 1 through Day 14 or Day 28 (depending on Cohort)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stoner, MD, Study Director — Rhythm Pharmaceuticals, Inc.